CLINICAL TRIAL: NCT04890860
Title: Detection of Right Ventricular Dysfunction by Portal Vein Doppler After Cardiac Surgery
Acronym: DVDDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020/08
Record Dates: First submitted 2021-05-03; First posted 2021-05-18 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2021-06

CONDITIONS: Postoperative Complications; Heart Diseases; Heart Failure; Heart Valve Diseases
Keywords: Cardiac surgery; Echocardiography; Right ventricular dysfunction; Doppler; Portal vein Doppler; Ventricular function
MeSH Terms: conditions — Postoperative Complications; Heart Diseases; Heart Failure; Heart Valve Diseases; Ventricular Dysfunction, Right

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults patients undergoing mitral and / or tricuspid valve surgery with cardiopulmonary bypass. (Experimental)
  Interventions: Other: cardiac surgery involving mitral or tricuspid valve repair procedure, with cardiopulmonary bypass

INTERVENTIONS:
Other: cardiac surgery involving mitral or tricuspid valve repair procedure, with cardiopulmonary bypass — cardiac surgery involving mitral or tricuspid valve repair procedure, with cardiopulmonary bypass

SUMMARY:
Right ventricular (RV) failure after cardiac surgery is associated with morbidity and mortality, but is hard to diagnose with conventional echocardiographic means. RV dysfunction may be associated with hepatic congestion, which may have an effect on portal veinous flow, but this has not been extensively. The investigators aimed determine whether an increased pulsatility in the portal venous flow was associated with RV dysfunction, after cardiac surgery at risk of RV dysfunction: mitral and tricuspid valve procedures.

DETAILED DESCRIPTION:
In cardiac surgical patients, RV dysfunction is associated with organ hypoperfusion and venous congestion leading to increased morbidity and mortality.

Non-invasive methods used to assess RV function are 2D-echocardiographic measurement of tricuspid annular plane systolic excursion (TAPSE), RV ejection fraction (EF), RV fractional area change (FAC), 3D assessment of RV function, tissue Doppler assessment of velocities, and magnetic resonance imaging (MRI). Though MRI is the gold standard method to assess RV function, it cannot be used in the perioperative period.

In the present prospective observational study, The investigators investigated the association between the pattern of portal venous flow and RV function as assessed by echocardiography in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old
* Ability to provide an informed consent
* Planned mitral and / or tricuspid valve surgery under cardiopulmonary bypass.

Exclusion Criteria:

* Insufficient echogenicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Right ventricular failure | First 24 hours post cardiac surgery
  1. systolic dysfunction (TAPSE below 16 mm or S wave below 9.5 cm/s)
  2. RV fractional area change below 35%
  3. End-diastole diameter ratio between RV and left ventricle > 0.6
  4. Ratio between S and D wave or inverse D wave in supra-hepatic veins
Portal flow measured by Doppler | First 24 hours post cardiac surgery
  flow pulsatility is assessed with the formula = 100 x (Vmax-Vmin)/Vmax. Time frame: First 24 hours post cardiac surgery

SECONDARY OUTCOMES:
Echocardiographic acquisition | First 24 hours post cardiac surgery
  Feasability of all measurements (RV failure with the 4 criteria:
  1. systolic dysfunction (TAPSE below 16 mm or S wave below 9.5 cm/s)
  2. RV fractional area change below 35%
  3. End-diastole diameter ratio between RV and left ventricle > 0.6
  4. Ratio between S and D wave or inverse D wave in supra-hepatic veins)
Echocardiographic acquisition | First 24 hours post cardiac surgery
  Feasability of all measurements (RV failure with the portal flow with Doppler)
Concordance of pulsatile flow assessment | First 24 hours post cardiac surgery
  Concordance of repeated measurements of the venous portal flow Time frame: First 24 hours post cardiac surgery
Concordance of RV dysfunction measurements | First 24 hours post cardiac surgery
  Concordance of repeated measurements of :
  1. systolic dysfunction (TAPSE below 16 mm or S wave below 9.5 cm/s)
  2. RV fractional area change below 35%
  3. End-diastole diameter ratio between RV and left ventricle > 0.6
  4. Ratio between S and D wave or inverse D wave in supra-hepatic veins
Preoperative RV dysfunction | 30 days before cardiac surgery
  As defined
  1. systolic dysfunction (TAPSE below 16 mm or S wave below 9.5 cm/s)
  2. RV fractional area change below 35%
  3. End-diastole diameter ratio between RV and left ventricle > 0.6
  4. Ratio between S and D wave or inverse D wave in supra-hepatic veins
Acute kidney injury | one week after surgery
  defined by KDIGO criteria as creatininemia elevation above > 26 micromol/L during the first 48 hours or +50% during the first week, oliguria with urine output less than 0.5 mL/kg/h during 6 hours.
Cholestasis | one week after surgery
  Conjugate bilirubin elevation above 12 mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- CMC Ambroise Paré, Neuilly-sur-Seine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haddad F, Couture P, Tousignant C, Denault AY. The right ventricle in cardiac surgery, a perioperative perspective: II. Pathophysiology, clinical importance, and management. Anesth Analg. 2009 Feb;108(2):422-33. doi: 10.1213/ane.0b013e31818d8b92. PMID 19151265
- [Background] Haddad F, Couture P, Tousignant C, Denault AY. The right ventricle in cardiac surgery, a perioperative perspective: I. Anatomy, physiology, and assessment. Anesth Analg. 2009 Feb;108(2):407-21. doi: 10.1213/ane.0b013e31818f8623. PMID 19151264
- [Background] Denault AY, Beaubien-Souligny W, Elmi-Sarabi M, Eljaiek R, El-Hamamsy I, Lamarche Y, Chronopoulos A, Lambert J, Bouchard J, Desjardins G. Clinical Significance of Portal Hypertension Diagnosed With Bedside Ultrasound After Cardiac Surgery. Anesth Analg. 2017 Apr;124(4):1109-1115. doi: 10.1213/ANE.0000000000001812. PMID 28151822
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859